CLINICAL TRIAL: NCT04453020
Title: Pilot Study to Evaluate Deep Brain Stimulation (DBS) of the Lateral Hypothalamic Area (LHA) on Energy Balance and Feeding Behavior in Patients With Chronic Refractory Obesity
Brief Title: Deep Brain Stimulation Effects in Patients With Chronic Refractory Obesity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The advent of GLP-1 medications for obesity has hampered successful recruitment. No subjects were consented nor enrolled into this study since the start date.
Sponsor: donald whiting (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor-Investigator, donald whiting, Principal Investigator, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Organization: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Obesity IDE
Record Dates: First submitted 2020-06-16; First posted 2020-07-01 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Obesity
Keywords: Deep Brain Stimulation; Lateral Hypothalamic Area; Feeding Behaviors; Energy Balance
MeSH Terms: conditions — Obesity; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- LHA DBS (Experimental): Subjects will receive bilateral DBS of the LHA
  Interventions: Device: DBS of the LHA

INTERVENTIONS:
Device: DBS of the LHA — Deep Brain Stimulation of the Lateral Hypothalamic Area
  Other Names: Vercise Gevia™ Deep Brain Stimulator System; Suretek Model DB-4600-C; Vercise Cartesia Directional Leads Model DB-2202-45; OR Cable and Extension Model DB-4100A; 8 Contact Extension Model NM-3138-55; Vercise Charging System Model DB-64125-US; Vercise Gevia 16 Contact IPG Kit Model DB-1200-S; Vercise DBS Remote Control 3 Kit Model DB-5552-1

SUMMARY:
This is a pilot study to evaluate the safety and efficacy of deep brain stimulation (DBS) of the lateral hypothalamic area (LHA) as a treatment for chronic refractory obesity. This study will include 6 individuals with chronic refractory obesity, that have failed other treatments including gastric bypass surgery.

DETAILED DESCRIPTION:
Six (N = 6) subjects with chronic refractory obesity will receive bilateral DBS implants in the LHA using the Boston Scientific Vercise Gevia DBS system. The primary objective is to evaluate the safety of DBS of the LHA using the current-driven Boston Scientific device and compare that to the safety data for our previous pilot using the voltage-driven DBS system for the treatment of chronic refractory obesity. The primary efficacy objective is to determine if DBS of the LHA can affect energy balance (i.e. energy intake and/or energy expenditure) in these patients. Secondary outcomes include quality of life outcomes and changes in feeding behaviors. Study participants will undergo a two-part DBS implantation procedure for placement of DBS electrodes in the LHA. Following this procedure, subjects with complete resting metabolic rate (RMR) testing to determine the optimal settings for the LHA stimulation. If effective, DBS technology might offer severely obese adults (BMI of ≥50 kg/m2), who have failed traditional therapy, a non-destructive, adaptable, reversible neurosurgical option for altering eating habits leading to sustained weight loss in the long-term.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients age ≥ 22 years and < 65 years old with a BMI of ≥ 40 kg/m2.
2. Failure of bariatric surgery (gastric bypass) and subjects who have no endoscopically or surgically correctable causes for failed bariatric surgery. "Failed bariatric surgery" is determined using the modified Reinhold classification as patients who are currently more than 50% over ideal body weight at least 24 months after a technically successful surgery (as confirmed by a esophagogastroduodenoscopy (EGD) within the 6 months prior to ICF).
3. Stable at their present weight (+/- 3 kg) for a 12-month period.
4. Neuropsychiatric evaluation must not reveal any issues that will be an impediment to subject's participation (as listed in Exclusion Criteria 2, 3 and 4).
5. Karnofsky Performance Score >60.
6. Platelet count >125,000 per cubic mm.
7. Prothrombin time (PT) and partial thromboplastin time (PTT) within normal limits.

Exclusion Criteria:

1. Any intracranial abnormality or medical condition that would contraindicate DBS surgery.
2. Have a history that includes a prior suicide attempt.
3. Have any significant psychiatric condition likely to compromise the subject's ability to comply with requirements of the study protocol (e.g. bipolar, schizophrenia, mood disorder with psychotic features, cluster B personality disorders) or have any prior history of schizophrenia or bipolar disorder or active psychotic episodes.
4. Have a current diagnosis of major depressive episode per DSM-IV (Diagnostics and Statistical Manual of Mental Disorders) criteria or has a current BDI-II score ≥ 17.
5. Any current drug or alcohol abuse, per DSM-IV criteria or any history of substance abuse (alcohol or other drug) or dependence during the past 12 months.
6. Any history of recurrent or unprovoked seizures.
7. Any history of hemorrhagic stroke.
8. Any diagnosis of acute myocardial infarction or cardiac arrest within previous 6 months.
9. Any diagnosis of a neurological disorder, such as multiple sclerosis, stroke, Parkinson's disease, severe brain atrophy or the presence of subdural hygromas or subdural hematomas.
10. Any history of hypothyroidism.
11. Any history of demonstrated binge eating.
12. Concurrent use of weight-loss prescription drug therapy or the use of over-the-counter weight loss preparations.
13. Any prior intracranial surgery or device implantation.
14. Any other active implanted devices (e.g., spinal cord stimulator, cochlear implant, pacemaker, vagus nerve stimulator) and /or drug delivery pumps, whether turned on or off. Passive implants (e.g., knee prostheses) would be allowed provided that they would not interfere with the DBS.
15. Any previously implanted Vagus Nerve Stimulation (VNS) patients.
16. A condition requiring or likely to require the use of Magnetic Resonance Imaging (MRI), diathermy or electroconvulsive therapy (ECT).
17. Likely to require the use of monopolar cautery, radio-frequency (RF) procedures, external defibrillation, lithotripsy, radiation therapy or transcranial stimulation.
18. Currently on any anticoagulant medications that cannot be discontinued during perioperative period.
19. Have any significant medical condition that is likely to interfere with study procedures or likely to confound evaluation of study endpoints, (e.g. hepatitis or HIV).
20. Any terminal illness with life expectancy of < 1 year.
21. Any diagnosis of malignancy (except basal cell of skin) within the past five years.
22. Any unresolved infection, a coagulopathy or significant cardiac or other medical risk factor for surgery.
23. Current or future risk of being immunocompromised (due to medications, disease factors, illness, etc.) that might significantly increase risk of infection.
24. Participation in any other clinical trial (e.g. drug, device, or biologics) concurrently or within the preceding 30 days. Participation in any other study will be allowed per investigator/sponsor discretion only.
25. Plan to receive any procedure that involves sudden jerking motions of the head or neck (e.g. certain chiropractic therapies) or massage and manipulation directly over the leads in the scalp, neck or chest, at any time during the study.
26. A female who is breastfeeding or of child-bearing potential with a positive urine pregnancy test or not using adequate contraception.
27. Not able to speak, write and read in English language as determined by the investigator.
28. Overall intellectual abilities below a standard score of 80 based on results from the Wechsler Abbreviated Scale of Intelligence (WASI; Wechsler, 1999)
29. Unable to fit into MRI or CT (Maximum weight limit is 180 kg (396 lb.).
30. Plasma pre-albumin < 14 mg/dL
31. Obesity as part of another medical condition, neurological injury or lesions, related to medication side effect, or as part of a genetic syndrome (i.e. Prader-Willi Syndrome, Leptin deficiency, etc.)
32. Be eligible for bariatric surgery revision including gastric outlet exclusion, gastrogastric fistula or other reasons that would qualify for a revision of their gastric bypass
33. Unable or unwilling to follow up for scheduled clinic visits

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Safety - Complication Rates | 12 months
  Adverse Events

SECONDARY OUTCOMES:
Resting metabolic rate (RMR) | Baseline, 2 months, 4-5 months and 20 months post-surgery
  RMR assessment of energy expenditure
Energy intake | 2 months and 4-5 months post-surgery
  Assessment of energy intake through ad libitum test meals
Impact of weight on quality of life: IWQOL-Lite | Baseline, 2 months and 4-5 months post-surgery
  Impact of Weight on Quality of Life Questionnaire (IWQOL-Lite). [Feeding behavior assessment]. There are 31 items by which the subject will respond to statements under 5 domains. Responses include: Always true, Usually true, Sometimes true, Rarely true, and Never true. All responses are totaled for a final score. Scores range from 0 to 100, with 100 representing the best quality of life.
Binge Eating Scale (BES) | Baseline, 2 months and 4-5 months post-surgery
  Eating Habits Checklist/Binge Eating Scale (BES). [Feeding behavior assessment]. There are 16 items that subjects will respond to. Each question has 3-4 separate responses assigned a numerical value. The score range is from 0-46. Higher scores equate to greater binging behavior.
Yale Food Addiction Scale | Baseline, 2 months and 4-5 months post-surgery
  Yale Food Addiction Scale. [Feeding behavior assessment]. There are 25 self-reported questions in dichotomous and Likert-type format. Food addiction is recognized when a subject meets at least three of the symptom criteria. The more symptoms met, the more severe the food addiction.
Power of Food Scale | Baseline, 2 months and 4-5 months post-surgery
  Power of Food Scale. [Feeding behavior assessment]. There are 21 items that subjects will assign a response to. The scale is as follows: 1=I don't agree at all, 2=I agree a little, 3=I agree somewhat, 4=I agree, 5=I strongly agree. All items are scored so that a higher item score indicates a greater responsiveness to the food environment.
Eating inventory | Baseline, 2 months and 4-5 months post-surgery
  Eating Inventory (EI). [Feeding behavior assessment]. There are 51 items consisting of three subscales. Scores range from a minimum of 0-0-0 to a maximum of 21-16-14. Higher scores are indicative of a greater level of the eating habits for the respective subscales.
Body shape perception | Baseline, 2 months and 4-5 months post-surgery
  Body Shape Questionnaire (BSQ). [Feeding behavior assessment]. There are 34 items that subjects will assign a response to. The scale is as follows: 1=Never, 2=Rarely, 3=Sometimes, 4=Often, 5=Very Often, 6=Always. The maximum score is 204, and a higher score indicates more dissatisfaction and discomfort with the body experience.
Food craving inventory | Baseline, 2 months and 4-5 months post-surgery
  Food Craving Inventory. [Feeding behavior assessment]. For each of the foods listed (37), subjects will rate the frequency of cravings. The scale is as follows: A=Never, B=Rarely (once or twice), C=Sometimes, D=Often, E=Always/almost every day. Cravings are measured for five types of foods. A total score is also obtained that measures the general construct of food cravings. Higher scores are indicative of more intense cravings.
Food preferences | Baseline, 2 months and 4-5 months post-surgery
  Food Preference Questionnaire. [Feeding behavior assessment]. Subjects rate their liking of 62 individual foods on a 5-point Likert scale. The scale is as follows: 1=Dislike a lot, 2=Dislike a little, 3=Neither like nor dislike, 4=Like a little, 5=Like a lot. Higher scores indicate a higher preference.
Delayed reward discounting | Baseline, 2 months and 4-5 months post-surgery
  Monetary Choice Questionnaire. [Feeding behavior assessment]. There are 21 items that subjects will indicate a response. The scale is as follows: 0=smaller reward today, 1=larger reward in the specified number of days. The questionnaire is scored by calculating where the respondent's answers place them amid reference discounting curves, where placement amid steeper curves indicates higher levels of impulsivity.
Appetitive sensations | Baseline, 2 months and 4-5 months post-surgery
  Visual analog scale (VAS) assessment. [Feeding behavior assessment]. Subjects will rank appetitive sensations on a scale from 0-10.
Quality of life measure: SF-36 | Baseline, 2 months and 4-5 months post-surgery
  Short Form-36 (SF-36). Subjects will rate responses to each of 36 items, (Likert and yes/no responses). Scores for each scale range from 0-100. The lower the score the more disability.
Depression score | Baseline, 2 months and 4-5 months post-surgery
  Beck Depression Inventory (BDI-II). There are 21 items where subjects will rate their responses on a Likert scale from 0-3. Total scores range from 0-63. Higher total scores indicate more severe depressive symptoms.
Changes in metabolic hormone profiles | 2 months and 4-5 months post-surgery
  Biochemical battery of tests. Blood draw for GLP1, PYY, Ghrelin (total and active) - Fasting
Body mass index | Baseline, 2 weeks, 2 months, 4-5 months, 6 months, 9 months, 12 months, 15 months, 18 months, 20 months and 24 months post-surgery
  Body Mass Index (BMI)
Change in DXA body composition | 2 months and 4-5 months post-surgery
  Change in body composition. Measured by dual-energy x-ray absorptiometry (DXA) scan

CONTACTS AND LOCATIONS:
Overall Officials: Donald Whiting, MD, Principal Investigator — Allegheny Health Network
Locations (1):
- Allegheny General Hospital, Pittsburgh, Pennsylvania, United States